CLINICAL TRIAL: NCT02021565
Title: Evaluating the CG ASSIST Program for Caregiving Dyads
Acronym: CG ASSIST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: D7873-R; 00050313 (Other: Emory IRB)
Record Dates: First submitted 2013-12-12; First posted 2013-12-27 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Transfer Impairment
Keywords: Caregivers; Activities of Daily Living; Dementia; Veterans; Self-Help Devices; Telemedicine
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: This study was a wait list control design. Participating couples were either assigned to the intervention group and received the full CG ASSIST program (assessment, observation, recommendations, equipment, modifications, and training) or were assigned to the delayed intervention control group (assessment and observation only). Then, as the intervention group was evaluated, the delayed intervention control group received the full CG ASSIST program. Both groups received 3-month follow-up observations and assessments. Results are reported for Baseline to T1 Intervention and Control.
Who Masked: Outcomes Assessor
Masking Description: The objective outcomes assessor did not know whether the participants were in the intervention or control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Receives the in-home training intervention immediately after completing the baseline assessment.
  The intervention includes three home visits from an AT Specialist (Occupational or Physical Therapist) who observes the dyad perform three ADL transfers, provides recommendations, equipment, home modifications, training, and follow-up training as needed.
  Interventions: Behavioral: Immediate Intervention Group
- Delayed Intervention Control Group (Other): Receives the in-home training intervention six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  Interventions: Other: Delayed Intervention Control Group

INTERVENTIONS:
Behavioral: Immediate Intervention Group — Assistive Technology (AT) Specialists, experts on assistive technology devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend assistive technology equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
  Other Names: In-home Training and Provision of AT (prn)
  Arms: Immediate Intervention Group
Other: Delayed Intervention Control Group — Receives the in-home training intervention six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  Other Names: Delayed In-home Training and Provision of AT (prn)
  Arms: Delayed Intervention Control Group

SUMMARY:
The CG ASSIST Project is a four-year study for older Veterans with transfer impairments and informal caregivers. CG ASSIST is an in-home training program for dyads designed to teach Veterans how to safely, skillfully, and (when possible) independently perform Activities of Daily Living involving transfers. Experts (OTs) who provide this training will also recommend, provide, and install assistive technology devices such as grab bars, bed rails, and toileting aids as needed. Research assistants conduct home visits with the dyads pre and post intervention to determine the effects of the program on Veteran and caregiver quality of life measures (burden, depression, task efficacy, lifespace).

Half of the couples in this study will receive the training from the expert remotely through a tele-video conferencing device. Research assistants will bring the device to participants' homes and assist in the training session.

DETAILED DESCRIPTION:
Introduction and Objective: The primary objective of the proposed four-year randomized, controlled trial is to document that providing a hands-on skills training and assistive technology (AT)/environmental modification program for older Veterans who are dependent in activities of daily living (ADLs) and their informal caregivers will result in improvements in caregiving processes (i.e., caregiving skills) and outcomes (i.e., safety during tasks) compared to the current standard of care and have beneficial direct and indirect effects for both members of the dyad. Secondary objectives are to determine the effects of the program on Veteran and caregiver subjective well-being (depression, quality of life) and to compare the relative effectiveness of two validated implementation modalities the traditional in-person approach and real-time interactive tele-video conferencing.

Research Plan. The study will be conducted with older Veterans (>60yrs) with mobility impairments who live in the community and are dependent on an informal caregiver for ADL assistance involving mobility, transfer or positional change. The study will utilize a modified randomized controlled cross-over design with four study arms and three or four outcome assessment periods. Prior to the first home visit, participants will be randomized to an intervention modality (in-person vs. tele-video) then randomized within those groups to an immediate intervention (IIG) or delayed intervention/control group (DICG).

Methods. In-home interviews will be completed with 180 Veteran caregiving dyads to obtain baseline, self-reported measures of caregiving needs, processes and outcomes using standardized, validated instruments. In-home visits by an Assistive Technology Specialist (ATS) will mirror the interview visits (within 1 week) to independently and objectively assess needs through observation of functional tasks. Dyads will be re-evaluated one (T2), two (T3), and four to five (T4) months later to ascertain change. Following T1 assessments, those in the IIG will receive 2 additional home visits from the ATS to (1) deliver the intervention and (2) reinforce the intervention. A 2nd blinded ATS will conduct the T2 outcome assessments. At T2 an ATS will conduct observation-based assessments which will also serve as a repeat baseline for the DICG. The intervention schedule will then be repeated for dyads in the DICG during T3. The final assessments for both groups will be collected 3 months after the intervention during T4.

Intervention. The Caregiver Assessment of Skill Sets & Individualized Support Thru Training or CG ASSIST program has recently undergone feasibility testing in a VA RR&D pilot study.

The intervention consists of (a) provision of assistive technology (AT) and simple home modifications to facilitate ADLs and (b) dyad training on the appropriate use of the devices and proper task execution using standardized protocols individualized to the needs and preferences of the dyad and environmental features of the home.

Clinical Relevance. Supporting and assisting caregivers in providing care for Veterans to help them age in place has important implications for the VHA system and the safety, dignity and quality of life of the Veterans we serve.

ELIGIBILITY:
Inclusion Criteria:

* Veterans 60 who require assistance from the identified caregiver with more than one Activity of Daily Living or three or more Instrumental Activity of Daily Living,
* have a life expectancy of greater than or equal to six (6) months,
* have no plans for transitioning out of home or into hospice in the next six months,
* and have approval from the primary care provider to participate in the research.
* Caregivers must live with the Veteran, provide care four (4) or more days out of the week for at least 6 months,
* and obtain a negative mini-cog assessment. Caregivers can be any relation (spouse, child, sibling, friend, etc.) to the Veteran so long as the two are cohabitating.
* Caregiver can be any age.

Exclusion Criteria:

* Caregivers who have a positive screen with the Mini-Cog fail to demonstrate cognitive capacity to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia C Griffiths, PhD, Principal Investigator — Atlanta VA Medical and Rehab Center, Decatur, GA
Locations (1):
- Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December 2013 and ended June 2016. Potential Veterans and informal/family caregivers were identified through the Department of Veterans Affairs Corporate Data Warehouse. The study was also advertised at community events and in local newspapers.
Groups:
- Immediate Intervention Group: Receives the in-home training intervention in-person immediately after completing the baseline assessment.
  In-home Training and Provision of Assistive Technology (prn): Assistive Technology (AT) Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Delayed Intervention Control Group: Receives the in-home training intervention in-person six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  In-home Training and Provision of Assistive Technology (AT) (prn): AT Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
Period: Baseline Through Intervention
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group
Started | 72 | 54
Caregivers | 36 | 27
Care Recipients | 36 | 27
Completed | 60 | 36
Not Completed | 12 | 18
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 8 | 8
Not completed — Protocol Violation | 0 | 7
Not completed — Lost to Follow-up | 4 | 2
Period: 3-month Follow-up
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group
Started | 60 | 36
Caregivers | 30 | 18
Care Recipients | 30 | 18
Completed | 50 | 34
Not Completed | 10 | 2
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Protocol Violation | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Immediate Intervention Group: Receives the in-home training intervention immediately after completing the baseline assessment.
  In-home Training and Provision of Assistive Technology (prn): Assistive Technology Specialists (ATSs), experts on assistive technology devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform four activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, ATSs also recommend assistive technology equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, ATSs provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Delayed Intervention Control Group: Receives the in-home training intervention six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  In-home Training and Provision of Assistive Technology (prn): Assistive Technology Specialists (ATSs), experts on assistive technology devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform four activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, ATSs also recommend assistive technology equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, ATSs provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Total: Total of all reporting groups
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group | Total
Number analyzed (Participants) | 72 | 54 | 126
Age, Customized [Mean (Standard Deviation); unit: years] — Population: The overall number of baseline participants differs from the number of analyzed participants because this study involved dyads (couples/pairs). Immediate Intervention group=36 dyads (36 caregivers + 36 care recipients = 72 participants). Delayed Intervention Control group=27 dyads(27 caregivers + 27 care recipients = 54 participants).
  years
    Caregiver Age: number analyzed (Participants) | 36 | 27 | 63
    Caregiver Age | 66 (9.5) | 66 (9.1) | 66 (9.4)
    Care Recipient Age: number analyzed (Participants) | 36 | 27 | 63
    Care Recipient Age | 74.3 (10.1) | 77.2 (9.3) | 75.5 (9.8)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: There were 58 caregivers who responded (Of original 63, 1 refused to answer, 4 screen failed or withdrew before reporting age).
  There were 62 Veteran care recipients who responded (Of original 63, 1 refused to answer).
  Participants
    Female Caregivers: number analyzed (Participants) | 34 | 24 | 58
    Female Caregivers | 34 | 22 | 56
    Male Veterans: number analyzed (Participants) | 35 | 27 | 62
    Male Veterans | 34 | 27 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Immediate Intervention Group Two caregivers withdrew before completing the baseline survey. Four care recipients withdrew before completing the baseline survey.
  Delayed Intervention Control Group Two caregivers failed screening. Two care recipients failed screening and four withdrew before completing the baseline survey.
  Participants
    Caregiver: number analyzed (Participants) | 34 | 25 | 59
    Caregiver: American Indian or Alaska Native | 0 | 0 | 0
    Caregiver: Asian | 1 | 1 | 2
    Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Caregiver: Black or African American | 20 | 13 | 33
    Caregiver: White | 13 | 10 | 23
    Caregiver: More than one race | 0 | 0 | 0
    Caregiver: Unknown or Not Reported | 0 | 1 | 1
    Care Recipient: number analyzed (Participants) | 32 | 21 | 53
    Care Recipient: American Indian or Alaska Native | 0 | 0 | 0
    Care Recipient: Asian | 0 | 0 | 0
    Care Recipient: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Care Recipient: Black or African American | 19 | 10 | 29
    Care Recipient: White | 13 | 11 | 24
    Care Recipient: More than one race | 0 | 0 | 0
    Care Recipient: Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72 | 54 | 126
Number of CG Health Problems [Mean (Standard Deviation); unit: Health problems] — Self-reported number of health problems reported by caregivers. Population: There were 35 caregivers assigned to the Immediate Intervention Group, but one withdrew before completing the baseline surveys.
  There were 28 caregivers assigned to the Delayed Intervention Control Group, but two failed the screening after consenting and one withdrew before completing the baseline surveys.
  Health problems
    number analyzed (Participants) | 34 | 25 | 59
    (all) | 2.47 (1.88) | 2.24 (1.63) | 2.37 (1.78)
Care Recipient Total Diagnoses [Mean (Standard Deviation); unit: Health Problems] — Population: Only the number of care recipients' health problems were summed from medical records. Caregiver health was self-reported
  Health Problems
    number analyzed (Participants) | 36 | 27 | 63
    (all) | 18.94 (9.86) | 23.33 (12.17) | 20.83 (11.12)
Marital Status [Count of Participants; unit: Participants] — Caregiver marital status (% married) Population: There were 36 caregivers assigned to the Immediate Intervention Group, but two withdrew before completing the baseline surveys.
  There were 27 caregivers assigned to the Delayed Intervention Control Group, but two failed the screening after consenting.
  Participants
    number analyzed (Participants) | 34 | 25 | 59
    (all) | 32 | 21 | 53
Education [Count of Participants; unit: Participants] — Caregiver education level (% education beyond high school) Population: Immediate Intervention Group One caregiver withdrew. One care recipient refused to answer and four withdrew.
  Delayed Intervention Control Group Two caregivers failed the screening and one withdrew. Two care recipients failed the screening and three withdrew.
  Participants
    Caregivers: number analyzed (Participants) | 34 | 25 | 59
    Caregivers | 22 | 18 | 40
    Care Recipients: number analyzed (Participants) | 32 | 22 | 54
    Care Recipients | 21 | 17 | 38
Employment [Count of Participants; unit: Participants] — Not employed is disabled or unable to work, unemployed, or never employed outside the home.
  Employed is part-time or full-time employment Population: Immediate Intervention Group One caregiver withdrew. One care recipient refused to answer and three withdrew.
  Delayed Intervention Control Group Two caregivers failed the screening and one withdrew. Two care recipients failed the screening and three withdrew.
  Participants
    Caregivers: number analyzed (Participants) | 34 | 25 | 59
    Caregivers: Retired | 20 | 14 | 34
    Caregivers: Not Employed | 11 | 8 | 19
    Caregivers: Employed | 3 | 3 | 6
    Care Recipients: number analyzed (Participants) | 32 | 22 | 54
    Care Recipients: Retired | 12 | 3 | 15
    Care Recipients: Not Employed | 6 | 7 | 13
    Care Recipients: Employed | 14 | 12 | 26
Income [Count of Participants; unit: Participants] — Caregiver reported income (% < 30,000) Population: There were 35 caregivers assigned to the Immediate Intervention Group, but one withdrew, four were unsure, and two refused to answer.
  There were 28 caregivers assigned to the Delayed Intervention Control Group, but two failed the screening after consenting, one withdrew, one was unsure, and two refused to answer.
  Participants
    number analyzed (Participants) | 28 | 22 | 50
    (all) | 11 | 10 | 21
Health Status [Count of Participants; unit: Participants] — Caregiver and care recipient self-reported health Population: Immediate Intervention Group One caregiver withdrew before completing the baseline surveys. Three care recipients withdrew. 17 care recipients did not respond (proxy).
  Delayed Intervention Control Group Two caregivers failed screening and three withdrew. Four care recipients withdrew, two failed screening, and 15 did not respond (proxy).
  Participants
    Caregivers: number analyzed (Participants) | 34 | 23 | 57
    Caregivers: Excellent | 2 | 4 | 6
    Caregivers: Very Good | 9 | 10 | 19
    Caregivers: Good | 21 | 6 | 27
    Caregivers: Fair | 2 | 2 | 4
    Caregivers: Poor | 0 | 1 | 1
    Care Recipients: number analyzed (Participants) | 16 | 8 | 24
    Care Recipients: Excellent | 0 | 0 | 0
    Care Recipients: Very Good | 1 | 1 | 2
    Care Recipients: Good | 10 | 0 | 10
    Care Recipients: Fair | 4 | 5 | 9
    Care Recipients: Poor | 1 | 2 | 3
Caregiver Relationship to Veteran [Count of Participants; unit: Participants] — Population: Responses are only from caregivers. Two caregivers from the Immediate Intervention Control Group withdrew before completing baseline assessments.
  Two caregivers from the Delayed Intervention Control Group failed screening.
  Participants
    number analyzed (Participants) | 34 | 25 | 59
    Spouse | 29 | 20 | 49
    Daughter | 3 | 3 | 6
    Sister | 1 | 1 | 2
    Neice | 0 | 1 | 1
    Mother | 1 | 0 | 1
Military Branch [Count of Participants; unit: Participants] — Branch of military in which Veteran care recipient served Population: Immediate Intervention Control Group One Veteran refused to answer and three withdrew.
  Delayed Intervention Control Group Two Veterans failed screening and two withdrew.
  Participants
    number analyzed (Participants) | 32 | 23 | 55
    Army | 16 | 13 | 29
    Navy | 5 | 2 | 7
    Air Force | 8 | 5 | 13
    Marines | 3 | 2 | 5
    Coast Guard | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Transfer Efficacy
Description: Caregiver reported the level of confidence that Veteran care recipient can perform 10 activity of daily living tasks rated on scale of 1-10. Efficacy in task completion reported both with assistance from the informal caregiver and performed independently by the Veteran. Scores range from 10-100 with higher scores reflecting greater transfer efficacy.
Time Frame: T1 Baseline and T2 Post Intervention; 4-6 Weeks
Population: Caregivers who reported their Veteran care recipient performed transfer tasks with assistance from informal caregiver. Two caregivers from the Intervention group and four caregivers from the Control group did not complete T2 and their data was not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Delayed Intervention Control Group: Control group.
  Receives the in-home training intervention six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  In-home Training and Provision of Assistive Technology (prn): Assistive Technology Specialists (ATSs), experts on assistive technology devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform four activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, ATSs also recommend assistive technology equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, ATSs provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group
Number analyzed (Participants) | 34 | 23
units on a scale
  Task Efficacy with Assistance from Caregiver T1 | 76.41 (25.06) | 79.57 (21.46)
  Task Efficacy With Assistance from Caregiver T2 | 64.44 (33.53) | 67.17 (35.71)
  Task Efficacy Independently T1 | 45.00 (24.78) | 41.91 (24.14)
  Task Efficacy Independently T2 | 44.69 (28.25) | 32.87 (25.03)
Statistical Analysis 1: Comparison: Immediate Intervention Group vs Delayed Intervention Control Group; Analysis 1 is for the caregiver reported confidence that Veteran care recipient can perform 10 transfer tasks with assistance from the informal caregiver; Test type: Superiority; p = 0.973, ANOVA — alpha = 0.025; Repeated measures
Statistical Analysis 2: Comparison: Immediate Intervention Group vs Delayed Intervention Control Group; Analysis 2 is for the caregiver reported confidence that Veteran care recipient can perform 10 transfer tasks independently; Test type: Superiority — Alpha = .025; p = 0.223, ANOVA

2. Secondary Outcome: Veteran Task Efficacy
Description: Veteran care recipient reported confidence in the performance of 10 activity of daily living tasks rated on scale of 1-10. Items are assessed for efficacy with and without (independently) assistance provided from a caregiver. Scores range from 10-100 with higher scores reflecting greater task efficacy.
Time Frame: T1 baseline and T2 Post Intervention; 4-6 weeks
Population: Veteran care recipient reported efficacy in performing transfer tasks with assistance from informal caregiver and independently. One Veteran from the Intervention group did not complete T2 and their data were not analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group
Number analyzed (Participants) | 35 | 27
units on a scale
  Task Efficacy With Assistance from Caregiver T1 | 85.73 (6.06) | 79.13 (8.31)
  Task Efficacy With Assistance from Caregiver T2 | 85.53 (4.85) | 83.75 (6.65)
  Task Efficacy Independent T1 | 62.60 (12.65) | 58.37 (24.17)
  Task Efficacy Independent T2 | 74.06 (13.85) | 70.50 (14.89)
Statistical Analysis 1: Comparison: Immediate Intervention Group vs Delayed Intervention Control Group; Analysis 1 is for the Veteran care recipient reported task efficacy; Test type: Superiority; p = 0.547, ANOVA
Statistical Analysis 2: Comparison: Immediate Intervention Group; Analysis 2 is for the Veteran reported confidence that he/she can perform 10 transfer tasks independently; Test type: Superiority; p = 0.891, ANOVA

3. Secondary Outcome: Caregiver Burden
Description: Zarit Burden Interview Revised -indicating caregiver burden. Caregivers endorse 22 items using a 5-point scale. Response options range from 0 (Never) to 4 (Nearly Always). Higher scores reflect greater caregiver burden. Scores range from 0 to 88.
Time Frame: T1 Baseline and T2 Post Intervention; 4-6 Weeks
Population: Composite caregiver burden reported by informal caregiver. Ten caregivers from the Intervention group and seven caregivers from the Control group did not complete T2 and their data was not analyzed.
Measure: Mean (Standard Deviation); unit: units on Zarit Burden scale
Arm/Group | Immediate Intervention Group | Delayed Intervention Control Group
Number analyzed (Participants) | 26 | 20
units on Zarit Burden scale
  Caregiver Burden T1 | 28.06 (14.31) | 29.14 (12.28)
  Caregiver Burden T2 | 26.00 (12.45) | 27.14 (11.65)
Statistical Analysis 1: Comparison: Immediate Intervention Group vs Delayed Intervention Control Group; Test type: Superiority; p = 0.729, ANOVA

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected for the duration of the study--2.5 years--from December 2013 until the study ended in June 2016.
Description: Because care recipients were required to receive assistance with at least one transfer, the majority of care recipient participants were frail. Each serious event reported to the team was recorded and reviewed. Only two potential injury adverse events were determined to be related to the research study because the events involved equipment provided during the intervention. All deaths and hospitalizations were determined to be anticipated due to the frail population and unrelated to the study.
Groups:
- Immediate Intervention Group - In-person: Receives the in-home training intervention in-person immediately after completing the baseline assessment.
  In-home Training and Provision of Assistive Technology (AT) (prn): AT Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Delayed Intervention Control Group - In-person: Receives the in-home training intervention in-person six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  In-home Training and Provision of Assistive Technology (AT) (prn): AT Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Immediate Intervention Group - Tele Arm: Receives the in-home training intervention remotely via a tele-video conference immediately after completing the baseline assessment.
  In-home Training and Provision of Assistive Technology (AT) (prn): AT Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
- Delayed Intervention Control Group - Tele Arm: Receives the in-home training intervention remotely via a tele-video conference six weeks after completing the initial baseline assessment. This allows for a control comparison group while still providing the intervention to all participants.
  In-home Training and Provision of Assistive Technology (AT) (prn): AT Specialists, experts on AT devices and how to performing transfer tasks, train Veteran and caregiver dyads to safely, skillfully, and (when appropriate) independently perform three activities of daily living (ADLs): transferring in and out of bed, toileting, and bathing. During the baseline assessments, AT Specialists also recommend AT equipment (grab bars, bed rails, raised toilet seats, etc.), environmental modifications, adaptive methods, and energy conservation techniques. On the first day of the intervention, AT Specialists provide and install recommended equipment and train the dyad to complete the three ADLs using the recommended the modified methods.
Arm/Group | Immediate Intervention Group - In-person | Delayed Intervention Control Group - In-person | Immediate Intervention Group - Tele Arm | Delayed Intervention Control Group - Tele Arm
All-Cause Mortality (participants affected / at risk) | 3/38 | 1/30 | 0/34 | 0/24
Serious Adverse Events (participants affected / at risk) | 7/38 | 9/30 | 3/34 | 0/24
Other Adverse Events (participants affected / at risk) | 0/38 | 0/30 | 0/34 | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Intervention Group - In-person (N=38) | Delayed Intervention Control Group - In-person (N=30) | Immediate Intervention Group - Tele Arm (N=34) | Delayed Intervention Control Group - Tele Arm (N=24)
Hospitalization (General disorders) | 5 (6) | 7 (7) | 3 (3) | 0 (0) — Participants self-reported hospitalizations that occurred while the Veteran was enrolled in this program. One participant in the Immediate Intervention Group was hospitalized twice while enrolled. He subsequently withdrew from the study.
Potential for Injury (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Participant fell while using equipment provided by the study, or the equipment fell near the participant. No injuries were reported.
Death (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) — Participant died while enrolled in this study.

LIMITATIONS AND CAVEATS:
The small sample size led to decreased power to detect a difference in the outcomes of interest so results should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes